CLINICAL TRIAL: NCT06173713
Title: Multi-Center, Non-Controlled, Prospective Radiostereometric Analysis of Emphasys Hip Solutions
Brief Title: Emphasys Radiostereometric Analysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Radiostereometric Analysis Network (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023:099
Record Dates: First submitted 2023-12-06; First posted 2023-12-18 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Emphasys Hip Solutions (Other): Emphasys Acetabular Shell, Emphasys AOX Polyethylene Liner, Articul/eze 12/14 metal head and Emphasys fem. stem
  Interventions: Device: Emphasys Hip Solutions

INTERVENTIONS:
Device: Emphasys Hip Solutions — Emphasys Acetabular Shell, Emphasys AOX Polyethylene Liner, Articul/eze 12/14 metal head and Emphasys fem. stem

SUMMARY:
This study is designed as a prospective, multi-centre, non-randomized, non-controlled study. This study does not limit the procedures involved in the treatment of the subject as long as the protocol specified products are utilized.

The primary objective is to establish the mean superior cup migration of the Emphasys Shell and the mean inferior stem migration of the Emphasys Stem using model-based RSA over the first two years post-implantation. Additionally, the data from this study will be compared to historical Pinnacle Acetabular Shell data obtained in study DSJ_2018_02.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals requiring primary THA for a severely painful and/or disabled joint from osteoarthritis, traumatic arthritis, rheumatoid arthritis, or congenital hip dysplasia, AVN of the femoral head or acute traumatic fracture of the femoral head or neck.
2. Individuals who are able to speak, read and comprehend the informed patient consent document and willing and able to provide informed patient consent for participation in the study and have authorized the transfer of his/her information to DePuy Synthes.
3. Individuals who are willing and able to return for follow-up as specified by the study protocol.
4. Individuals who are a minimum age of 21 years at the time of consent.
5. Individuals who are willing and able to complete the Subject Hip Outcomes questionnaires as specified by the study protocol.

Exclusion Criteria:

1. Individuals who have active local or systemic infection.
2. Individuals who have loss of musculature, neuromuscular compromise or vascular compromise that would impact rehabilitation following surgery.
3. Individuals with poor bone quality, such as osteoporosis, where in the surgeon's opinion, there could be considerable migration of the prosthesis or require additional acetabular cup fixation using screws, or a significant chance of fracture of the femoral shaft and/or the lack of adequate bone to support the implant(s).
4. Individuals with Charcot's or Paget's disease.
5. Individuals who, in the judgement of the investigator, would not be a candidate for protocol allowable components to be used for their THA.
6. Women who are pregnant or lactating.
7. Individuals who have had a contralateral hip that was implanted less than 6 months prior to the time of consent into this study or individuals that expect to have a contralateral hip implanted in the following 6 months at the time of consent into this study.
8. Individuals that have amputations in either leg that would impact rehabilitation following surgery.
9. Individuals who are bedridden
10. Individuals that have participated in a clinical investigation with an investigational product (drug or device) in the last three months.
11. Individuals currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
12. Individuals, in the opinion of the Investigator, who are drug or alcohol abusers or have a psychological disorder that could affect their ability to complete patient reported questionnaires or be compliant with follow-up requirements.
13. Individuals diagnosed and taking prescription medications to treat a muscular disorder that limits mobility due to sever stiffness and pain such as fibromyalgia or polymyalgia.
14. Subject has a medical condition with less than 2 years life expectancy.
15. Individual has a BMI >45 kg/m2.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Migration - Shell | 2 Years
  The mean vertical subsidence (Y translation, also known as superior shell migration) at 2 years as measured with RSA.
Migration - Stem | 2 Years
  The mean vertical subsidence (Y translation, also known as inferior stem migration) at 2 years as measured with RSA.

SECONDARY OUTCOMES:
Subsidence - Emphasys Shell | 6 months, 1 Year
  RSA measured subsidence of the Emphasys Shell at 6 months and 1 year and to compare it to historical Pinnacle Shell data
Subsidence - Emphasys Stem | 6 months, 1 Year
  RSA measured subsidence of the Emphasys Stemat 6 months and 1 year
Other RSA measurements - Emphasys Shell | 6 Weeks, 6 months, 1 year and 2 years
  Other RSA measurements of the Emphasys Shell (X and Z translations in mm, X, Y, and Z rotations in degrees, and maximal total point motion in mm) at all time points. These endpoints will be compared to historical Pinnacle Shell data.
Other RSA measurements - Emphasys Stem | 6 Weeks, 6 months, 1 year and 2 years
  Other RSA measurements of the Emphasys Stem (X and Z translations in mm, X, Y, and Z rotations in degrees, and maximal total point motion in mm) at all time points. These endpoints will be compared to historical Pinnacle Shell data.
Head Penetration (in mm) | 1 year and 2 years
  Linear head penetration (in mm) at 1 year and 2 years. This endpoint will be compared to historical Pinnacle data.
HOOS Jr. | Pre-op, 6 weeks, 6 months, 1 year and 2 years
  Functional and health status will be measured with HOOS Jr. This is a patient-reported outcome measure for which scores range from 0 to 100; a score of 0 indicating total hip disability and 100 indicating optimal hip health.These endpoints will be compared to historical Pinnacle data.
Harris Hip Score | Pre-op, 6 weeks, 6 months, 1 year and 2 years
  Functional score will be measured with Harris Hip Score. The score has a maximum of 100 points (best possible outcome) covering pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points). These endpoints will be compared to historical Pinnacle data.
Forgotten Joint Score (FJS-12) | Pre-op, 6 weeks, 6 months, 1 year and 2 years
  Functional and health status will be measured with the Forgotten Joint Score (FJS-12). The FJS total score range is 0-100, higher scores indicating the patient is able to forget the joint daily lower degree of joint awareness. These endpoints will be compared to historical Pinnacle data.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Turgeon, MD, Principal Investigator — Concordia Hospital
Locations (1):
- Orthopaedic Innovation Centre, Winnipeg, Manitoba, Canada